CLINICAL TRIAL: NCT05370430
Title: A Phase 1 Study Evaluating BAFFR-targeting CAR T Cells for Patients With Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma (B-NHL)
Brief Title: BAFFR-targeting CAR T Cells for Patients With Relapsed or Refractory B-NHL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PeproMene Bio, Inc. (Industry)
Collaborators: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMB-102; PMB-BAFFR-102 (Other: PeproMeneBio)
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma
Keywords: Relapsed or Refractory; Mantle Cell Lymphoma; BAFFR-CAR T cells; B-cell Non-Hodgkin's Lymphoma; B-NHL; BAFFR; MCL; LBCL
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell; Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- B-cell activating factor receptor-Chimeric antigen receptor T cells [BAFFR-CAR T cells] (Experimental): BAFFR-CAR T cells in participants with r/r B-NHL
  Interventions: Biological: BAFFR-CAR T cells

INTERVENTIONS:
Biological: BAFFR-CAR T cells — First-in-human trial examining the safety and preliminary efficacy of BAFFR-CAR T cells in participants with r/r B-NHL

SUMMARY:
A Phase 1 Study Evaluating BAFFR-targeting CAR T Cells for Patients with Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma (B-NHL)

DETAILED DESCRIPTION:
This phase I trial evaluates the side effects and best dose of BAFFR-CAR T cells in treating patients with B-cell Non-Hodgkin's Lymphoma (B-NHL) that has come back (recurrent) or does not respond to treatment (refractory). T cells are infection fighting blood cells that can kill cancer cells. The T cells given in this study will come from the patient and will have a new gene put in them that makes them able to recognize BAFFR, a protein on the surface of cancer cells. These BAFFR-specific T cells may help the body's immune system identify and kill BAFFR+ cancer cells.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent: Signed informed consent by the participant or legally authorized representative.
2. Age & Performance Status:

   * Age ≥ 18 years
   * ECOG performance status ≤ 2
3. Diagnosis & Disease Criteria:

   * Histologically confirmed B-NHL, including LBCL, MCL, and FL/MZL subtypes meeting specified prior treatment conditions.
   * BAFF-R expression on lymphoma cells required.
4. Measurable Disease: Tumor ≥1.5 cm on CT/PET scan or evidence of disease in blood, BM, GI, skin, or spleen.
5. Prior CAR T-cell Therapy: Allowed if ≥ 3 months since last treatment and CD19 CAR-T persistence < 5% before leukapheresis.
6. Organ Function & Laboratory Criteria:

   * Hematologic: ANC ≥ 1000/μL, Platelets ≥ 75,000/μL (exceptions for BM involvement).
   * Liver Function: Bilirubin ≤ 1.5x ULN (except Gilbert's), AST/ALT < 3x ULN.
   * Renal Function: CrCl ≥ 50 mL/min.
   * Cardiac & Pulmonary: LVEF ≥ 45%, QTcF ≤ 480 ms, O₂ saturation > 91% on room air.
7. Infectious Disease Screening: Seronegative for HIV, active HBV, active HCV (or undetectable viral load if positive).
8. Reproductive Considerations:

   * Negative pregnancy test for females of childbearing potential.
   * Use of effective contraception or abstinence through 3 months post-treatment.

Exclusion Criteria:

1. Prior Therapies & Transplants:

   * Prior allogeneic SCT.
   * Autologous SCT < 6 months before leukapheresis.
   * Concurrent systemic steroids or chronic immunosuppressant use.
2. Disease-Specific Exclusions:

   * Cardiac lymphoma involvement.
   * Need for urgent therapy due to tumor-related complications (e.g., bowel obstruction).
3. Medical Conditions:

   * Active autoimmune disease requiring immunosuppressants.
   * Primary immunodeficiency.
   * Cardiac conditions, including NYHA Class III/IV heart disease, arrhythmia, recent MI (≤ 6 months), stroke (≤ 6 months), or significant VTE (≤ 6 months).
   * Neurologic conditions, including prior optic neuritis, CNS inflammatory diseases, or seizure disorders.
   * History of malignancy, unless resected/treated with curative intent or in remission for ≥ 3 years.
   * Uncontrolled systemic infections or active CNS lymphoma.
4. Pregnancy & Breastfeeding: Females who are pregnant or nursing.
5. Other Considerations:

   * Investigator-determined safety concerns.
   * Potential noncompliance with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2027-07-13 (Estimated); Study Completion 2028-06-13 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 1 year post treatment
  Assess the safety of administering BAFFR-CAR T cells in participants with relapsed or refractory (r/r) B-cell Non-Hodgkin's Lymphoma (B-NHL) and it's subtypes. Toxicity will be graded per Common Terminology Criteria for Adverse Events version 5.0, Cytokine Release Syndrome (CRS) and neurotoxicity which use the American Society for Transplantation and Cellular Therapy Consensus Criteria (ASTCT) and Graft versus Host Disease (GVHD) criteria. Toxicities will be followed from the start of lymphodepletion until the end of the study.
Maximum Tolerated Dose (MTD) | The DLT evaluation period is defined as 28 days following BAFFR CAR-T infusion.
  Determine the maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D) of BAFFR-CAR T cells. The highest dose with ≤ 1/6 participants with DLT will be considered the MTD.

SECONDARY OUTCOMES:
Disease Response | Up to 1 year post treatment
  Defined as achieving a best response of complete response or partial response per Lugano Criteria
Minimal Residual Disease (MRD) | Up to 1 year post treatment
  Negative MRD is defined by malignant cells < 0.01% by flow cytometry or clonoSEQ.
B Cell Quantification | Up to 1 year post treatment
  Measured by flow cytometry
Progression-free survival (PFS) | From CAR T cell infusion to the first observation of disease relapse/progression or death from any cause, whichever occurs first, assessed up to 15 years.
  Kaplan-Meier product limit method with log-log transformation for the confidence interval will be used to estimate PFS.
Overall Survival (OS) | From the day of BAFFR-CAR T cell infusion to death from any cause assessed, up to 15 years.
  Kaplan-Meier product limit method with log-log transformation for the confidence interval will be used to estimate OS.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Budde, MD, Study Chair — City of Hope Medical Center
Locations (6):
- United States (6):
  - City of Hope Medical Center, Duarte, California
  - Stanford University, Stanford, California
  - University of Kansas Hospital, Kansas City, Kansas
  - University of Minnesota, Minneapolis, Minnesota
  - Atrium Health Levine Cancer Institute - Morehead, Charlotte, North Carolina
  - Providence Swedish Cancer Institute, Seattle, Washington

REFERENCES:
- [Derived] Dong Z, Budde LE, Oh E, Szymura S, Anderson A, Del Real M, Cha SC, Forman SJ, Kwak LW, Wang X. Analysis of polyfunctionality for enhanced BAFF-R CAR T-cell therapy for hematologic malignancies. Blood Adv. 2024 Aug 13;8(15):4066-4076. doi: 10.1182/bloodadvances.2024013195. PMID 38885481